CLINICAL TRIAL: NCT06995534
Title: Comparison of Static Hand-Wrist Splinting and Exercise Therapy in the Management of De Quervain's Tenosynovitis
Brief Title: Splinting vs Exercise in De Quervain's Tenosynovitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Konya Beyhekim Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, eda ünal madıoğlu, doctor, Konya Beyhekim Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KonyaBeyhekimTRH2023/4689
Record Dates: First submitted 2025-05-12; First posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Splints; Exercise Therapy; De Quervains Tenosynovitis; Pain Management; Ultrasonographic
Keywords: pain; De Quervains Tenosynovitis; exercise therapy; splints; Ultrasonographic
MeSH Terms: conditions — De Quervain Disease; Agnosia; Pain | interventions — Splints; Exercise Therapy

STUDY DESIGN:
Intervention Model Description: Other: Static Wrist-Hand Resting Splint (Thumb Spica Splint) Other: Exercise Therapy
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Static Hand-Wrist Splinting (Other)
  Interventions: Other: splint
- Exercise Therapy (Other)
  Interventions: Other: Exercise Therapy

INTERVENTIONS:
Other: splint — static wrist-hand splint + education on activity modification and positioning in daily life
  Arms: Static Hand-Wrist Splinting
Other: Exercise Therapy — Home-based Exercise Therapy + Education on activity modification and positioning in daily life
  Arms: Exercise Therapy

SUMMARY:
De Quervain's disease is a painful tenosynovitis of the abductor pollicis longus and extensor pollicis brevis muscle tendons located in the first dorsal compartment. The primary treatment for De Quervain's disease is conservative; surgical intervention is rarely required. Currently, there is no standardized treatment protocol supported by strong, up-to-date evidence.

The aim of this study is to compare the effectiveness of a static hand-wrist resting splint and exercise therapy in the conservative treatment of De Quervain's tenosynovitis. Patients will be evaluated in terms of pain levels, functional/symptom status, hand-finger strength, pressure pain threshold (PPT), tendon cross-sectional area measured by ultrasound, and the presence of effusion findings (semiquantitative; 0-3), and patient satisfaction.

DETAILED DESCRIPTION:
Patients who meet the inclusion and exclusion criteria will undergo a detailed clinical examination and medical history review, after which written informed consent will be obtained. They will then be randomly assigned to one of the two treatment groups using block randomization.

Baseline sociodemographic data (age, sex, body mass index, employment status, education level, marital status) and clinical variables (dominant hand, symptom duration, comorbidities, affected hand, presence of the Finkelstein sign, pain severity, functional/symptom status, hand-finger strength, pressure pain threshold (PPT), and ultrasonographic findings) will be recorded.

Patients in the first group will be provided with a static wrist-hand resting splint with thumb support, extending to the distal forearm. They will be instructed to wear the splint for at least 6-8 hours per day for a minimum of 4 weeks. Additionally, both groups will receive training on activity modification and positioning.

Patients in the second group will be given a home exercise program. They will perform the exercises twice daily for 6 weeks, with each exercise consisting of 10 repetitions. All patients will be evaluated at baseline, at the second week of treatment, and at the end of the sixth week.

Outcome measures will include clinical examination findings (Finkelstein test), pain severity [Visual Analog Scale (VAS) at rest and during activity], the Turkish versions of the Disabilities of the Arm, Shoulder and Hand (DASH) Questionnaire, Health Assessment Questionnaire (HAQ), and Patient-Rated Wrist Evaluation (PRWE), patient satisfaction, handgrip and finger pinch strength measurements, and pain pressure threshold using an algometer.

Ultrasound evaluations of the abductor pollicis longus and extensor pollicis brevis tendons in the first dorsal compartment including the measurement of the cross-sectional area (csa) will be performed at baseline, week 2, and week 6.

All assessments will be conducted by the same blinded investigator who is unaware of the group allocations

ELIGIBILITY:
Inclusion Criteria:

* Adults aged between 18 and 65 years

Patients experiencing wrist pain and tenderness for less than 3 months and clinically diagnosed with acute or subacute De Quervain's tenosynovitis

Visual Analog Scale (VAS) pain score ≥ 3

Exclusion Criteria:

* History of trauma

Wrist fractures

Local infection

Presence of rheumatologic diseases (e.g., rheumatoid arthritis, psoriatic arthritis)

Presence of symptomatic hand osteoarthritis

Continuous use of nonsteroidal anti-inflammatory drugs (NSAIDs) or corticosteroids

Receipt of physical therapy for the hand or wrist within the past 3 months

Corticosteroid injection into the hand or wrist within the past 3 months

Diagnosed with significant neurological disorders (e.g., upper motor neuron disease)

Presence of uncontrolled systemic diseases (e.g., uncontrolled diabetes mellitus, congestive heart failure, chronic kidney disease, hepatic failure)

Major psychiatric disorders

Communication difficulties

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
VAS pain | baseline, week 2 and week 6
  VAS pain activity and rest: 0 no pain; 10 unbearable/max. pain.
Patient Rated Wrist Evaluation( PRWE) | baseline, week 2 and week 6
  The Patient-Rated Wrist Evaluation (PRWE) is a brief and effective self-report questionnaire that allows patients to assess their own wrist and hand problems. The PRWE consists of two main subscales: the Pain Subscale (0-50 points) and the Function Subscale (0-50 points). The total score ranges from 0 (no disability) to 100 (maximum pain and functional impairment).
The Disabilities of the Arm, Shoulder and Hand (DASH) | baseline, week 2 and week 6
  The Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire is a self-reported outcome measure used to assess the impact of upper extremity disorders on daily activities. It consists of 30 items, each scored on a 5-point Likert scale ranging from 1 (no difficulty) to 5 (unable to perform). The total score ranges from 0 to 100, where 0 indicates no disability and 100 indicates severe functional limitation.

SECONDARY OUTCOMES:
Hand grip strength | baseline, week 2 and week 6
  Hand Grip Strength (HGS):
  Following the definitions outlined in the literature, HGS will be measured using Jamar hand dynamometers. The patients will be asked to squeeze the dynamometer three times with maximum strength, allowing 30-60 seconds of rest between each attempt. The average force (in pounds/kg) will then be recorded.
Finger pinch strength | baseline, week 2 and week 6
  Finger Pinch Strength (FGS):
  Following the definitions outlined in the literature, FGS will be measured using Baseline pinch dynamometers. The patients will be asked to squeeze the dynamometer three times with maximum strength, allowing 30-60 seconds of rest between each attempt. The average force (in pounds/kg) will then be recorded.
Ultrasonographic evaluation of the first dorsal compartment tendons | Baseline, week 2 and week 6
  Ultrasonographic evaluation of the Abductor Pollicis Longus (APL) Extensor Pollicis Brevis (EPB) will be performed with a LA2-14A transducer /superficial linear probe(Samsung).The patient is seated with the forearm in a neutral position and the palm resting on a flat surface. The wrist is slightly extended to expose the radial side. A high-frequency linear transducer (typically 10-18 MHz) is placed transversely over the radiocarpal joint at the wrist, just proximal to the radial styloid.
  The first dorsal compartment is visualized in cross-sectional (short axis) view. Both tendons (APL and EPB) appear as oval or round hyperechoic structures within the tendon sheath. Peritendinous edema is assessed semiquantitatively (0-3based on its visual appearance around the tendon.CSA (mm2) measurements will be performed using USG with high sensitivity, reflecting tendon thickening or swelling due to inflammation. The mean of three measurements will be calculated for analysis.
Patient satisfaction | week 2 and week 6
  Patient satisfaction (Subjective impression of improvement):
  Satisfaction levels of patients will be questioned. In the assessment consisting of five clauses with Likert-type scales, the clauses will be described as follows: 1, 'no satisfaction at all'; 2, 'no satisfaction'; 3, neutral (no positive or negative effect); 4, 'satisfied'; and 5, 'very satisfied'.

CONTACTS AND LOCATIONS:
Locations (1):
- Konya Beyhekim Training and Research Hospital, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No